CLINICAL TRIAL: NCT01163825
Title: An Open Label, Dose-Escalation Study of Encapsulated Cell Biodelivery of Nerve Growth Factor to the Cholinergic Basal Forebrain of Alzheimer´s Disease Patients
Brief Title: Encapsulated Cell Biodelivery of Nerve Growth Factor to Alzheimer´s Disease Patients
Acronym: NsG0202
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NsGene A/S (Industry)
Collaborators: Karolinska Institutet (Other); Region Stockholm (Other Government)
Responsible Party: Lars U. Wahlberg, MD, PhD, Exec.VP, COO, CMO, NsGene A/S
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NsG0202-001
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Nerve Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nerve Growth Factor (Experimental): Dose 1
  Interventions: Drug: Nerve Growth Factor
- Nerve Growth Factor 2 (Experimental): Dose 2
  Interventions: Drug: Nerve Growth Factor

INTERVENTIONS:
Drug: Nerve Growth Factor — Encapsulated cell biodelivery of Nerve Growth Factor (NGF) to the basal forebrain nuclei of the brain by multiple implantable devices housing NGF-secreting human cells

SUMMARY:
Cholinergic neurons in the basal forebrain project widely to the cerebral cortex and hippocampus. These neurons depend on nerve growth factor (NGF) from their target areas for survival. Impaired NGF supply is part of the Alzheimer's disease (AD) pathology, and the degeneration of these neurons correlates with the cognitive decline in these patients. The objective of encapsulated cell biodelivery (ECB) is to maintain normal levels of NGF to support cholinergic function. NsGene's NGF secreting ECB device (NsG0202) combines the potential benefits of targeted gene therapy with the safety of a retrievable implantable device.

The study is an open label, single centre, 12-month, dose-escalation phase Ib study in patients with mild to moderate AD. The primary objective is safety and tolerability, while secondary outcomes measure include cognition, behaviour, neuropsychology, activities of daily living (ADL), positron emission tomography (PET) imaging and electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years
2. All patients must fulfil the NINDNDS-ARDRA criteria of Alzheimer's disease.
3. The subject must have a score between 15-24 inclusive, on the mini-mental state examination (MMSE).
4. The subject must have a caregiver who is able and committed to assist the subject to comply with the trial protocol, and who is willing to provide the information required at assessment interviews.
5. Informed consent must be obtained from the subject together with a close caregiver, in accordance with the requirements of the ethical committee.

Exclusion Criteria:

1. A diagnosis of Schizophrenia, Schizo-affective disorder or paranoid disorder according to DSM IV without any suspicion cognitive decline.
2. Patients with the following co-existing medical conditions:
3. History of seizures.
4. Brain tumor including meningeoma.
5. Clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances.
6. Clinically significant back pain.
7. Bleeding disorders.
8. Patients who, in the opinion of the investigator, are otherwise unsuitable for a trial of this type.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 12 months

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) | 12 months
  Cognition using ADAS-Cog, neuropsychologic test battery

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Jönhagen, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Machado A, Ferreira D, Grothe MJ, Eyjolfsdottir H, Almqvist PM, Cavallin L, Lind G, Linderoth B, Seiger A, Teipel S, Wahlberg LU, Wahlund LO, Westman E, Eriksdotter M; Alzheimer's Disease Neuroimaging Initiative. The cholinergic system in subtypes of Alzheimer's disease: an in vivo longitudinal MRI study. Alzheimers Res Ther. 2020 May 6;12(1):51. doi: 10.1186/s13195-020-00620-7. PMID 32375872
- [Derived] Eyjolfsdottir H, Eriksdotter M, Linderoth B, Lind G, Juliusson B, Kusk P, Almkvist O, Andreasen N, Blennow K, Ferreira D, Westman E, Nennesmo I, Karami A, Darreh-Shori T, Kadir A, Nordberg A, Sundstrom E, Wahlund LO, Wall A, Wiberg M, Winblad B, Seiger A, Wahlberg L, Almqvist P. Targeted delivery of nerve growth factor to the cholinergic basal forebrain of Alzheimer's disease patients: application of a second-generation encapsulated cell biodelivery device. Alzheimers Res Ther. 2016 Jul 7;8(1):30. doi: 10.1186/s13195-016-0195-9. PMID 27389402
- [Derived] Wahlberg LU, Lind G, Almqvist PM, Kusk P, Tornoe J, Juliusson B, Soderman M, Sellden E, Seiger A, Eriksdotter-Jonhagen M, Linderoth B. Targeted delivery of nerve growth factor via encapsulated cell biodelivery in Alzheimer disease: a technology platform for restorative neurosurgery. J Neurosurg. 2012 Aug;117(2):340-7. doi: 10.3171/2012.2.JNS11714. Epub 2012 Jun 1. PMID 22655593